CLINICAL TRIAL: NCT06792318
Title: Use of Fibroblast Activation Protein Inhibitor (FAPI) PET-CT Before Surgery in Patient with Endometriosis
Brief Title: The Role of FAPI PET-CT in Diagnosing Endometriosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, Israel Sandler, MD, Ziv Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 101-24-ZIV; IRB Number 101-24-ZIV (Other: Ziv Medical Center, Safed)
Record Dates: First submitted 2025-01-15; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Endometriosis
Keywords: endometriosis; PET CT; Fibroblast activation protein inhibitor
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: All participants undergo FAPI PET-CT imaging followed by laparoscopic surgery. Surgical specimens are sent for pathological confirmation of PET-CT findings. This single-group diagnostic study aims to evaluate the accuracy of FAPI PET-CT in detecting endometriosis lesions using surgical and pathological findings as the gold standard.
Masking Description: Open label study. The surgeon operates based on PET-CT findings, and the pathologist examines specimens from lesions detected on PET-CT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FAPI PET-CT Diagnostic Arm (Experimental): Participants undergo FAPI PET-CT imaging at multiple timepoints (10, 30, 60, and 80 minutes post-injection) using a single FAPI dose. Each participant will then undergo laparoscopic surgery with tissue sampling for pathological confirmation of endometriotic lesions.
  Interventions: Diagnostic Test: FAPI PET-CT

INTERVENTIONS:
Diagnostic Test: FAPI PET-CT — FAPI PET-CT imaging protocol:
  Single dose 68Ga/18F-FAPI (2 MBq/kg)
  Two imaging sessions:
  First: 10 and 30 minutes post-injection Second: 60 and 80 minutes post-injection Ultra-low dose CT for attenuation correction and anatomical localization

SUMMARY:
Patients with suspected endometriosis scheduled for surgery will be identified. They will be asked to participate in a study evaluating the feasibility of FAPI PET-CT in diagnosing endometriosis. The results will be compared with surgical findings, pathology, and other imaging techniques if available (i.e., MRI, US).

DETAILED DESCRIPTION:
This study investigates FAPI PET-CT imaging in endometriosis diagnosis using a standardized protocol. Participants will undergo two imaging sessions after a single FAPI injection:

First Session:

Initial scan at 10 minutes post-injection Follow-up scan at 30 minutes

Second Session:

Additional scans at 60 and 80 minutes post-injection

The protocol is designed to minimize radiation exposure through:

Single FAPI injection Two ultra-low dose CT scans Limited field of view to suspected areas. Nuclear medicine physicians will review PET-CT images independently, blinded to other imaging findings (MRI, US). Results will be shared with surgeons to guide the removal of suspicious lesions during surgery. All removed tissue will undergo pathological examination for confirmation.

The study incorporates safety monitoring:

Observation during and after FAPI administration Follow-up contact at 24-48 hours post-scan Documentation of any adverse events Immediate reporting of unexpected findings. This research could potentially provide evidence for a novel, non-invasive method to comprehensively map endometriotic lesions, improving pre-operative planning.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18-45 years
* Clinical suspicion of endometriosis based on symptoms
* Scheduled for diagnostic/therapeutic laparoscopic surgery
* Ability to understand and provide written informed consent
* Completed and signed Radiation Exposure Documentation Form

Exclusion Criteria:

* Pregnant women or women who are breastfeeding
* History of pelvic radiation therapy
* Known active malignancy
* Exposure to ionizing radiation for medical purposes within 12 months prior to enrollment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of FAPI PET-CT in Endometriosis Detection | Within 1 month post-surgery
  Assessment of FAPI PET-CT diagnostic performance through calculation of sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV). Surgical findings with histological confirmation will serve as the reference standard for evaluation.

SECONDARY OUTCOMES:
Comparison of FAPI PET-CT with Conventional Imaging | Within 1 month post-surgery
  Evaluation of FAPI PET-CT's ability to detect endometriotic lesions not visible on conventional imaging (TVUS and MRI). Comparison includes identification of additional lesions and assessment of anatomical distribution of detected lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv Medical Center, Safed, Israel

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in published articles will be shared after deidentification. Data will be available beginning 9 months and ending 36 months following article publication. Data will be shared with researchers who provide a methodologically sound scientific proposal. Proposals should be directed to [israels@ziv.gov.il]. Data requestors will need to sign a data access agreement. Data will include deidentified participant data related to FAPI PET-CT findings and surgical/pathological outcomes.
Supporting Information: Study Protocol, SAP
Time Frame: Start: "9 months after publication" End: "36 months following publication"
Access Criteria: Qualified researchers can submit a proposal to access de-identified IPD and supporting documents. The proposal should include: research objectives, statistical analysis plan, research team qualifications, and funding source. Upon approval, researchers must sign a data access agreement. Data will be shared via a secure institutional platform.

REFERENCES:
- [Background] Zhao L, Kang F, Pang Y, Fang J, Sun L, Wu H, Lan X, Wang J, Chen H. Fibroblast Activation Protein Inhibitor Tracers and Their Preclinical, Translational, and Clinical Status in China. J Nucl Med. 2024 May 6;65(Suppl 1):4S-11S. doi: 10.2967/jnumed.123.266983. PMID 38719234
- [Background] Fox R, Chang S, Hicks L, Mooney S, Rogers PAW, Hicks RJ, Tyson K, Holdsworth-Carson SJ. Positron emission tomography in the evaluation of endometriosis: A systematic review. Eur J Obstet Gynecol Reprod Biol. 2024 Aug;299:258-265. doi: 10.1016/j.ejogrb.2024.06.017. Epub 2024 Jun 12. PMID 38917749
- [Background] Garcia Garcia JM, Vannuzzi V, Donati C, Bernacchioni C, Bruni P, Petraglia F. Endometriosis: Cellular and Molecular Mechanisms Leading to Fibrosis. Reprod Sci. 2023 May;30(5):1453-1461. doi: 10.1007/s43032-022-01083-x. Epub 2022 Oct 26. PMID 36289173
- [Background] Pascoal E, Wessels JM, Aas-Eng MK, Abrao MS, Condous G, Jurkovic D, Espada M, Exacoustos C, Ferrero S, Guerriero S, Hudelist G, Malzoni M, Reid S, Tang S, Tomassetti C, Singh SS, Van den Bosch T, Leonardi M. Strengths and limitations of diagnostic tools for endometriosis and relevance in diagnostic test accuracy research. Ultrasound Obstet Gynecol. 2022 Sep;60(3):309-327. doi: 10.1002/uog.24892. PMID 35229963
- [Background] Parasar P, Ozcan P, Terry KL. Endometriosis: Epidemiology, Diagnosis and Clinical Management. Curr Obstet Gynecol Rep. 2017 Mar;6(1):34-41. doi: 10.1007/s13669-017-0187-1. Epub 2017 Jan 27. PMID 29276652